CLINICAL TRIAL: NCT01742013
Title: Randomized, Double-blinded, Placebo-controlled, Multicenter Investigator Initiated Clinical Study to Explore the Efficacy and Safety of GCJBP Laennec Inj.(Human Placenta Hydrolysate) 4ml Per Day 3 Times Per Week for 6 Weeks in the Chronic Fatigue Patients With Chronic Fatigue Syndrome or Idiopathic Chronic Fatigue
Brief Title: Investigator Initiated Clinical Study to Explore the Efficacy and Safety of Human Placenta Hydrolysate in the Chronic Fatigue Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ho Cheol Shin, M.D., Ph.D. (Other)
Collaborators: Ajou University School of Medicine (Other); Green Cross Corporation (Industry); Symyoo (Industry)
Responsible Party: Sponsor-Investigator, Ho Cheol Shin, M.D., Ph.D., Professor, Kangbuk Samsung Hospital
Organization: Kangbuk Samsung Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Laennec-IIT
Record Dates: First submitted 2012-11-29; First posted 2012-12-05 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Fatigue Syndrome; Idiopathic Chronic Fatigue
Keywords: Chronic Fatigue; CFS; ICF; human placenta
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): NaCl 0.9%, s.c., 4ml (2ml x 2), 3 times per a week, 6 weeks
  Interventions: Drug: Placebo
- GCJBP Laennec Inj. (Experimental): GCJBP Laennec Injection,s.c., 4ml(2ml x 2)/day, 3 times per a week, 6 weeks
  Interventions: Drug: GCJBP Laennec Inj.

INTERVENTIONS:
Drug: GCJBP Laennec Inj. — Test drug
  Other Names: Human placenta hydrolysate
  Arms: GCJBP Laennec Inj.
Drug: Placebo — Comparator
  Other Names: Normal saline solution (NaCl 0.9%)
  Arms: Placebo

SUMMARY:
GCJBP Laennec Injection contains a variety of cytokines derived from human placenta, amino acids, peptides, nucleobases, and carbohydrates. This product is approved for improving liver function. Also, it has been prescribed for lots of diseases such as menopausal disorders, atopic dermatitis, skin cares as well as fatigue for long time. Although its action mechanism and clinical effectiveness are not still clear, there are reports which say a strong probability of its clinical effectiveness in the chronic fatigue patients.

This study aims to investigate the safety and efficacy of GCJBP Laennec Inj. (Human placenta hydrolysate) in the chronic fatigue patients through a randomized controlled tial.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with chronic fatigue syndrome or idiopathic chronic fatigue
* Given written informed consent
* Male or female aged between 20 and 65
* Patient who can read and answer to written questionnaires
* Patient who agrees to visit clinic for study drug injection 3 times per a week for 6 weeks

Exclusion Criteria:

* Patient who has been administrated with any other investigational product for 28 days prior to screening visit
* Patient who is pregnant or childbearing potential female patient who does not consent for contraception during the study
* Patient who has a hypersensitivity provoked by study drug or others drived from animals
* Patient who has been received with any human placenta product for 6 months before study participation
* Abnormal liver function
* Abnormal renal function
* Back Depression Inventory (BDI) II is more than 29
* Underlying disease/conditions, in the investigator's judgment, which will be unable to participate in the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change of Fatigue Severity Scale (FSS) | Baseline and 6 weeks

SECONDARY OUTCOMES:
Change per item of Fatigue Severity Scale (FSS) | Baseline, 3, 6 and 9 weeks
Rate of patients whose FSS decreased from 4 and more to less than 4 | Baseline, 3, 6 and 9 weeks
Change of Visual Analogue Scale (VAS) | Baseline, 3 and 6 weeks
Change of Multidimensional Fatigue Inventory (MFI) | Baseline, 3 and 6 weeks
Global Improvement Scale (GIS) | 6 weeks
  GIS assessment after 6-week study treatment by investigator
Change in the concentration of salivary cortisol | Baseline and 6 weeks
Change in the concentration of interleukin-6 and interleukin 1b | Baseline and 6 weeks
Heart Rate Variability (HRV) parameters at resting | Baseline and 6 weeks
Drug compliance | 6 weeks
  Compliance rate of used study drugs to prescribed study drugs after 6-week treatment
Adverse Events | 9 weeks
  All adverse events reported for study duration of 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheol Shin, M.D., Ph.d., Principal Investigator — Kangbuk Samsung Hospital
Locations (2):
- South Korea (2):
  - Kangbuk Samsung Hospital, Seoul
  - Ajou University Hospital, Suwon